CLINICAL TRIAL: NCT05717088
Title: Effectiveness of Oral Sucrose for Preterm Infants Undergoing Point-of-care Lung Ultrasound: A Randomized Controlled Trial
Brief Title: Effectiveness of Oral Sucrose During Lung Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 20-0220-E
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-01

CONDITIONS: Pain
Keywords: Preterm, Lung, PIPP score, infants, neonates
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The random numbers will be placed in sequentially numbered, sealed, opaque envelopes and will be opened after obtaining informed consent and just before the procedure by one of the study investigators to ensure allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral sucrose + soother group (group A) (Experimental): Group A: Infants will receive oral sucrose (24%) followed by a soother 2 minutes before the procedure "LUS scan". The dose will be 0.2 mL, 0.5 mL and 1 mL for infants with current weight < 1500g, 1500-2500g, and > 2500g respectively.
  Interventions: Other: 24% Sucrose solution
- Soother alone group (group B) (No Intervention): Group B (control group): infants will receive a soother 2 minutes before LUS scan.

INTERVENTIONS:
Other: 24% Sucrose solution — Infants will either receive oral sucrose (24%) 2 minutes before the procedure "LUS scan". The dose will be 0.2 mL, 0.5 mL and 1 mL for infants with current weight < 1500g, 1500-2500g, and > 2500g respectively.
  Arms: Oral sucrose + soother group (group A)

SUMMARY:
Background: control of pain in neonates has an important role in preventing long- term effects on neurodevelopment and pain reactivity. Oral sucrose and non-nutritive suckling are considered a non-pharmacological treatment that has many advantages. Currently, there is controversy regarding the use of sucrose during point of care lung ultrasound (LUS) scan as many consider LUS is not a painful procedure.

Objective: Determine the efficacy of oral sucrose solution + soother versus soother alone in reducing infant's agitation during LUS scan Method: This is a blinded, prospective, parallel group randomized controlled trial comparing the Premature infant pain profile (PIPP) score in infants randomized to receive oral sucrose followed by soother soother vs. soother alone while having LUS scan Study outcomes: The primary outcome of this study is to compare the changes in PIPP scores at 4 time points between infants receiving oral sucrose solution + soother versus soother alone. The secondary outcomes are 1) total time to complete a standard LUS scan from start of scanning to the end, 2) Association of LUS with adverse events e.g., episodes of desaturation, tachycardia, bradycardia or apnea.

DETAILED DESCRIPTION:
Hypothesis: The investigators hypothesize that oral sucrose solution with soother is more effective than soother alone in reducing infant's agitation during LUS.

Method

Design: This is a prospective randomized controlled trial comparing PIPP score during LUS in infants who receive oral sucrose plus soother vs. soother alone.

Population: described below

Intervention The study is a 2-arm, randomized controlled trial. Infants will be allocated to one of the 2 groups as described below

Study Procedures:

Infants' face and physiological monitor will be video recorded for 30 seconds before administration of study intervention. Video recording will be paused during the administration of study intervention (24% sucrose + soother or soother alone) to be given while maintaining blinding of type of intervention and group assignment for enrolled infants. Video recording will be restarted after administration of the study intervention and will be continued for 1 minute after finishing the scan and returning the baby to pre-intervention state. In infants assigned to group A, the study solution (24% oral sucrose) will be given by a study investigator or bedside nurse to the anterior portion of the tongue without touching the infant's mouth followed by insertion of a soother that will be maintained in infant's mouth throughout the procedure. Infants assigned to group B will receive a soother that will be maintained in infant's mouth throughout the procedure. PIPP score will be assessed at 4-time points a) 30 seconds prior to administration of study intervention (baseline PIPP score), b) 30 seconds into LUS scan, c) midway of LUS scan, d) 30 seconds after the procedure is completed and soother removed.

Outcome measures: The primary and secondary outcomes as described below

Measures Measurement of procedural pain For all enrolled infants, The investigators will assess stress/pain using PIPP score, a validated tool approved by the American Academy of Pediatrics for pain assessment in both term and preterm neonates. The PIPP score is based on seven parameters: corrected gestational age, behavioral state, changes in maximum heart rate (HR), changes in minimum arterial oxygen saturation (SpO2), brow bulging, eye squeezing, and nasolabial furrowing. These indices are individually scored from 0 to 3, and the total score is calculated by summing the scores for these 7 indices. The PIPP score ranges from 0-21 in preterm infants.

Measurement of physiological response Heart rate (HR) and Oxygen saturation (SpO2) data will be videotaped directly from the patient's bedside physiological monitor (Philips-The intellivue MX800). HR and SpO2 will be reviewed by videotape analyzer and will be incorporated into PIPP score. Average HR and SpO2, presence of apnea during the LUS will reviewed and documented to assess for adverse events associated with the study procedure.

Measurement of incidence of adverse events The following adverse events associated with the procedure (LUS scan); tachycardia> 180 bpm, bradycardia< 100 bpm, SpO2 < 80%, or apnea (cessation of breathing for > 20 second or < 20 second but associated with hypoxia or bradycardia) will be compared between the 2 study groups.

Randomization, allocation and blinding All enrolled infants will be randomized by computer-generated randomization sequence (block size from 4 to 6 with 1:1 allocation ratio) to 24% sucrose plus soother group or soother alone (control group). The random numbers will be placed in sequentially numbered, sealed, opaque envelopes and will be opened after obtaining informed consent and just before the procedure by one of the study investigators to ensure allocation concealment. These envelopes will be kept in a secure, locked drawer in the principle investigator office and only study investigators will have access to it. Attending physician will be blinded, however, the operator who will perform the LUS will not be possible due to nature of intervention. The PIPP score analyzer (the coder) will be blind to group allocation.

Sample size The sample size is calculated based on the results of a previous study that assessed pain/stress associated with echocardiography in neonates using the Premature Infant Pain Profile (PIPP) score. The investigators hypothesize a difference of 2 or more in the mean PIPP score between the control and the intervention group. Assuming standard deviation of 2.5 for both groups, with 5% significance level and 80% power, 26 subjects are required in each group. The investigators are planning to recruit 32 subjects in each group (total 64) to account for 20% loss due to errors in videotaping and missing data.

Consent Parents/legal guardians of infants who meet eligibility criteria will be approached for participation in the study. One of the study investigators (who is not involved in infant's care at the time of the consent) will provide a brief description of the research and state clearly that participation is voluntary and that refusal would not change the care that the infant will receive in the unit. Parents/legal guardians who agree to participate will sign a written consent form.

Statistical Analysis Infant characteristics as well as outcomes will be compared between two groups. Difference will be assessed by Pearson Chi-square or Fisher exact test for categorical variables, and Student t-test (ANOVA F-test) or Wilcoxon rank test for continuous variables. Results will be reported as frequency (percentage), mean (standard deviation) or median (inter quartile range) as appropriate. GEE model will be used to assess the significance between two groups with repeat measures. All analyses will be conducted using SAS 9.4 (SAS Institute Inc., Cary, NC) with two-sided significance level 0.05.

Data collection The following data will be collected; Infants' baseline characteristics; gestational age(GA), Birth weight, sex, current/corrected GA and weight, APGAR score at 5 minutes) will be collected. Data regarding current respiratory support at the time of the study will be collected. Total time needed to complete a scan will abstracted from ultrasound machine. Adverse events during the scan such as tachycardia (> 180 bpm), bradycardia (< 100 bpm), Oxygen saturation (< 80%), or apnea episode will be recorded. All patients' identifiers will be removed. A separate list of study ID and Hospital ID (MSID) will be kept on secure hospital drive with password-protected access available only to study investigators.

ELIGIBILITY:
Inclusion Criteria: Patient must meet all inclusion criteria to be eligible for participation that include;

* Preterm infants (GA < 37 weeks) admitted to the neonatal intensive care unit, Mount Sinai Hospital,
* Undergoing LUS for clinical or research purpose,
* Hemodynamically stable (not requiring any circulatory support), and
* Written informed parental consent is obtained.

Exclusion Criteria:

* Infants with neurological disorders, congenital anomalies that interfere with oral intake,
* On pain medications, or
* receiving nothing per oral because of medical condition e.g. necrotizing enterocolitis are excluded

Ages: 0 Days to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Premature infant pain profile Score (PIPP) measured in (points 0-21) ranging 0-21 points | 1 YEAR
  To compare the changes in the Pain Score "Premature infant pain profile Score (PIPP)" at 4 time points between infants receiving oral sucrose solution + Pacifier versus Pacifier alone. PIPP score ranges from 0-21 points, where 0 means no pain and 21 is severe pain.

SECONDARY OUTCOMES:
Total time to complete the scan (minutes) | 1 YEAR
  1) total time to complete a standard LUS scan from start of scanning to the end, 2) Association of LUS with adverse events e.g., episodes of desaturation, tachycardia, bradycardia or apnea.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Mohamed, MD, Principal Investigator — Sinai Health System
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada